CLINICAL TRIAL: NCT05827497
Title: Baricitinib, Methotrexate as Monotherapy or Combination in the Treatment of Rheumatoid Arthritis - an Open Label Randomized Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Md. Abu Shahin, Professor of Rheumatology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2022/10476
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Rheumatoid Arthritis
Keywords: baricitinib, rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): baricitinib 2 mg once daily
  Interventions: Drug: Baricitinib 2 MG
- Group B (Active Comparator): methotrexate on 25 mg weekly
  Interventions: Drug: Methotrexate 25mg

INTERVENTIONS:
Drug: Baricitinib 2 MG — baricitinib 2 mg once daily
  Other Names: Baricitinib 2mg
  Arms: Group A
Drug: Methotrexate 25mg — 25mg daily
  Arms: Group B

SUMMARY:
The goal of this open-label randomized clinical trial is to assess the efficacy of baricitinib 2 mg in comparison to methotrexate 25 mg as monotherapy followed by baricitinib 4 mg in comparison to methotrexate 10 mg and baricitinib 2 mg combination in patients with rheumatoid arthritis with moderate to severe disease activity. The main question it aims to answer:

• Is there any difference in the efficacy of baricitinib as monotherapy in comparison to methotrexate monotherapy or methotrexate-baricitinib combination in the treatment of rheumatoid arthritis

DETAILED DESCRIPTION:
This open-label randomized clinical trial will be conducted in the department of rheumatology, BSMMU. The rheumatoid arthritis patients with moderate to high disease activity at baseline, disease activity score (DAS28ESR>3.2) will be considered as primary entry criteria for this study. Consecutive sampling method will be applied. The study will be done in 2 phases, duration of each phase 24 weeks. Considering inclusion and exclusion criteria, total 132 patients are randomized into group A and group B following block randomization. Each group will be consisting of 66 patients. In phase 1 Group A will be put on baricitinib 2 mg once daily and Group B will be put on methotrexate 25 mg weekly. The patients who fail to achieve remission or low disease activity by 24 weeks eligible for entry into phase 2 where group A will be put on baricitinib 4 mg and group B will be put on baricitinib 2 mg in combination with methotrexate 10 mg. Follow-up will be done at the 4th, 12th and 24th week in phase 1 and 28th, 36th and 48th week in phase 2. Response to treatment will be evaluated by DAS 28 ESR. At the end of 24th week endpoint for efficacy will be assessed at by DAS 28ESR. Adverse effects will be assessed by history, physical examinations and investigations.

Results will be compared among two groups with a 95% confidence interval and a p-value of < 0.05. The degrees of statistical significance between groups will be analyzed by unpaired t-test and/or Mann-Whitney U test. Qualitative data in between groups will be analyzed by the chi-square test. Probabilities of associations will be assessed by calculating Spearman´s rank correlation coefficient

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients more than 18 years of age 2. Patients fulfill the ACR/EULAR 2010 classification criteria for Rheumatoid arthritis 3. Patients with DAS 28 ESR> 3.2

Exclusion Criteria:

* 1. Recent or concurrent infection including active tuberculosis 2. Haemoglobin (Hb) < 9 gm/dl 3. Total WBC count < 4000 / µL 4. Neutrophil count < 1200 / µL 5. Lymphocyte count < 750 / µL 6. AST/ALT > three times the upper limit of normal 7. Estimated glomerular filtration rate < 60 ml/minute/1.73 m2 8. Co-morbid illness- e.g., Malignancy 9 . Pregnant or breast feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
DAS 28 ESR | 24 weeks
  Following parameters are used to evaluate DAS28- Tender joint count Swollen joint count Patient global assessment (vas in cm) ESR/CRP

SECONDARY OUTCOMES:
Clinical disease activity index (CDAI) | 24 weeks
  Tender joint count Swollen joint count Patient global assessment (vas in cm) Physician global assessment (vas in cm)
Health assessment questionnaire disability index (HAQ-DI) | 24 weeks
  The patient reports the amount of difficulty they have in performing some of these activities like Dressing and grooming, Arising, Eating, Walking, Hygiene, Reach, Grip and Activities. Each question asks on a scale ranging from 0 to 3. If the categories performed without any difficulty (scale 0) up to cannot be done at all (scale 3)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Md Abu Shahiin, FCPS, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Dr. Md. Abu Shahin, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleischmann R, Schiff M, van der Heijde D, Ramos-Remus C, Spindler A, Stanislav M, Zerbini CA, Gurbuz S, Dickson C, de Bono S, Schlichting D, Beattie S, Kuo WL, Rooney T, Macias W, Takeuchi T. Baricitinib, Methotrexate, or Combination in Patients With Rheumatoid Arthritis and No or Limited Prior Disease-Modifying Antirheumatic Drug Treatment. Arthritis Rheumatol. 2017 Mar;69(3):506-517. doi: 10.1002/art.39953. PMID 27723271
- [Background] Islam N, Baron Basak T, OudeVoshaar MA, Ferdous N, Rasker JJ, Atiqul Haq S. Cross-cultural adaptation and validation of a Bengali Health Assessment Questionnaire for use in rheumatoid arthritis patients. Int J Rheum Dis. 2013 Aug;16(4):413-7. doi: 10.1111/1756-185X.12032. Epub 2013 Jan 22. PMID 23992261
- [Background] Yamaoka K. Janus kinase inhibitors for rheumatoid arthritis. Curr Opin Chem Biol. 2016 Jun;32:29-33. doi: 10.1016/j.cbpa.2016.03.006. Epub 2016 Mar 17. PMID 26994322